CLINICAL TRIAL: NCT01157299
Title: Hemodynamic Evaluation of Preload Responsiveness in Children by Using PiCCO
Acronym: PreloaDren
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitario La Paz (Other)
Responsible Party: Pedro de la Oliva, Hospital Universitario La Paz
Other Study IDs: HULP-PI-800
Record Dates: First submitted 2010-07-06; First posted 2010-07-07 (Estimated); Last update posted 2010-07-07 (Estimated); Status verified 2010-06

CONDITIONS: Shock; Sepsis; Systemic Inflammatory Response Syndrome; Low Cardiac Output; Dilated Cardiomyopathy
Keywords: Hemodynamics; Pediatric Intensive Care Unit; Low cardiac output; Thermodilution; Stroke volume; Global end-diastolic volume; Fluid responsiveness; Passive leg raising; Infant
MeSH Terms: conditions — Shock; Sepsis; Systemic Inflammatory Response Syndrome; Cardiac Output, Low; Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Hemodynamic instability: Hypotension and/or evidence of end-organ hypoperfusion
- Hemodynamic stability: Normotension and end-organ normoperfusion along with
  * Vasopressor, vasodilator or inotropic therapy
  * Edema and/or evidence of hypervolemia
- Hemodinamically "normal": Normotension and end-organ normoperfusion along with
  * Non vasopressor, vasodilator or inotropic therapy
  * Normohydration state
  * Non Systemic Inflammatory Response Syndrome
  * Spontaneous breathing and PEEP, or CPAP, equal or less than 5 cm H2O

SUMMARY:
The purpose of this study is

* To assess the value of dynamics (SVV, PPV) and static indices (GEDVI, ITBVI, CVP) of preload and its combination with contractility (CI,SV, ventricular power, dP/dtmax, CFI, GEF) and lung water indices (ELWI), as predictors of fluid responsiveness in both spontaneously breathing and mechanically ventilated pediatric patients.
* To assess the value of stroke volume and pulse pressure changes from femoral pulse contour analysis (PiCCO2) during passive leg raising as predictor of fluid responsiveness in pediatric patients.
* To establish normal and cutoff values of transpulmonary thermodilution (PiCCO2) hemodynamic variables in hemodynamically stables and hemodynamically "normal" patients.

DETAILED DESCRIPTION:
One of the ongoing challenges in critical care has been determining adequate fluid resuscitation. Overly aggressive volume expansion may produce deleterious effects, especially in patients with respiratory, renal and/or cardiac failure. Since the clinical ability to judge hemodynamic parameters is known to be poor, the determination of variables that would predict response to fluid challenge would be important for clinical decision-making.

Traditional measures of preload (CVP, PAOP) are now known to be incapable to assess the volume status and fluid responsiveness, especially in children.

There are two kinds of reasons for explaining the failure of markers of preload to predict volume responsiveness: the first reason is that the markers commonly used at the bedside are not always accurate measures of cardiac preload; the second reason is that an assessment of preload is not an assessment of preload responsiveness.

The rapid determination of hemodynamic status offered by noninvasive hemodynamic devices as PICCO2 would allow tailoring of volume expansion necessary in hypoperfusion states to increase left ventricular volume and cardiac output. Studies in critically ill adults patients have demonstrated that passive leg raising autotransfusion and functional hemodynamic monitoring, by using pulse contour analysis, are reliable in the detection of fluid responsiveness. However, currently we have very few studies in pediatric patients using arterial pulse contour analysis and transpulmonary thermodilution, which does not allow the rational application of the hemodynamic variables for guiding fluid resuscitation.

This study pretend to assess 1) the value of dynamics and static indices of preload, and its combination with contractility and lung water indices, as predictors of fluid responsiveness in both spontaneously breathing and mechanically ventilated pediatric patients and 2) the value of stroke volume and pulse pressure changes during passive leg raising autotransfusion, as predictors of fluid responsiveness in pediatric patients.

In this observational study, the hemodynamical variables are registered during the hemodynamically unstable, stable and "normal" states of the pediatric patient and before and after clinically indicated fluid (crystalloid, colloid or hemoderivative) infusion. Passive leg raising hemodynamic changes will be compared with the hemodynamic changes caused by fluid infusion.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients admitted to PICU
* Patient equipped with a femoral arterial catheter and central venous catheter or who requires advanced hemodynamic monitoring
* Parents consent

Exclusion Criteria:

* Absolute

  * Patient with left to right cardiac shunts
  * Patient with extra-corporeal life support
  * Less than 4 Kg body weight
* For passive leg raising procedure

  * Patient with head trauma or intracranial hypertension
  * Patient in prone position
  * Patient who may not tolerate supine or Trendelenburg position: ej. Glenn procedure
  * Patient with hip injury

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients admitted to the PICU equipped with a femoral arterial catheter and a central venous catheter or who require advanced hemodinamic monitoring
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-08 (Estimated); Study Completion 2010-09 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Pedro de la Oliva, MD PhD., Study Director — Hospital Universitario La Paz; Ignacio Sánchez-Díaz, MD PhD, Principal Investigator — Hospital Universitario 12 de Octubre de Madrid; Elena Alvarez-Rojas, MD, Principal Investigator — Hospital Universitario Ramón y Cajal de Madrid; Susana Jaraba-Caballero, MD, Principal Investigator — Hospital Universitario Reina Sofia de Córdoba; Patricia Roselló-Millet, MD, Principal Investigator — Hospital Clínico Universitario de Valencia; José Manuel González-Gómez, MD, Principal Investigator — Hospital Universitario Carlos Haya de Málaga; Ana Serrano-Gonzalez, MD PhD, Principal Investigator — Hospital Infantil Universitario del Niño Jesús; Eduardo Consuegra-Llapur, MD, Principal Investigator — Hospital Universitario Materno-Infantil de las Palmas de Gran Canaria
Locations (7):
- Spain (7):
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Infantil Universitario del Niño Jesús, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Clinico Universitario, Valencia

REFERENCES:
- [Background] Brierley J, Carcillo JA, Choong K, Cornell T, Decaen A, Deymann A, Doctor A, Davis A, Duff J, Dugas MA, Duncan A, Evans B, Feldman J, Felmet K, Fisher G, Frankel L, Jeffries H, Greenwald B, Gutierrez J, Hall M, Han YY, Hanson J, Hazelzet J, Hernan L, Kiff J, Kissoon N, Kon A, Irazuzta J, Lin J, Lorts A, Mariscalco M, Mehta R, Nadel S, Nguyen T, Nicholson C, Peters M, Okhuysen-Cawley R, Poulton T, Relves M, Rodriguez A, Rozenfeld R, Schnitzler E, Shanley T, Kache S, Skippen P, Torres A, von Dessauer B, Weingarten J, Yeh T, Zaritsky A, Stojadinovic B, Zimmerman J, Zuckerberg A. Clinical practice parameters for hemodynamic support of pediatric and neonatal septic shock: 2007 update from the American College of Critical Care Medicine. Crit Care Med. 2009 Feb;37(2):666-88. doi: 10.1097/CCM.0b013e31819323c6. PMID 19325359
- [Background] Michard F, Descorps-Declere A, Lopes MR. Using pulse pressure variation in patients with acute respiratory distress syndrome. Crit Care Med. 2008 Oct;36(10):2946-8. doi: 10.1097/CCM.0b013e318187b6fd. No abstract available. PMID 18812805
- [Background] Osman D, Ridel C, Ray P, Monnet X, Anguel N, Richard C, Teboul JL. Cardiac filling pressures are not appropriate to predict hemodynamic response to volume challenge. Crit Care Med. 2007 Jan;35(1):64-8. doi: 10.1097/01.CCM.0000249851.94101.4F. PMID 17080001
- [Background] Lichtwarck-Aschoff M, Zeravik J, Pfeiffer UJ. Intrathoracic blood volume accurately reflects circulatory volume status in critically ill patients with mechanical ventilation. Intensive Care Med. 1992;18(3):142-7. doi: 10.1007/BF01709237. PMID 1644961
- [Background] Michard F, Alaya S, Zarka V, Bahloul M, Richard C, Teboul JL. Global end-diastolic volume as an indicator of cardiac preload in patients with septic shock. Chest. 2003 Nov;124(5):1900-8. doi: 10.1378/chest.124.5.1900. PMID 14605066
- [Background] Teboul JL, Monnet X. Prediction of volume responsiveness in critically ill patients with spontaneous breathing activity. Curr Opin Crit Care. 2008 Jun;14(3):334-9. doi: 10.1097/MCC.0b013e3282fd6e1e. PMID 18467896
- [Background] Monnet X, Teboul JL. Passive leg raising. Intensive Care Med. 2008 Apr;34(4):659-63. doi: 10.1007/s00134-008-0994-y. Epub 2008 Jan 23. PMID 18214429
- [Background] Heenen S, De Backer D, Vincent JL. How can the response to volume expansion in patients with spontaneous respiratory movements be predicted? Crit Care. 2006;10(4):R102. doi: 10.1186/cc4970. PMID 16846530
- [Background] Kim HK, Pinsky MR. Effect of tidal volume, sampling duration, and cardiac contractility on pulse pressure and stroke volume variation during positive-pressure ventilation. Crit Care Med. 2008 Oct;36(10):2858-62. doi: 10.1097/CCM.0b013e3181865aea. PMID 18766112
- [Background] Pinsky MR. Heart-lung interactions. Curr Opin Crit Care. 2007 Oct;13(5):528-31. doi: 10.1097/MCC.0b013e3282efad97. PMID 17762231
- [Background] Cecchetti C, Stoppa F, Vanacore N, Barbieri MA, Raucci U, Pasotti E, Tomasello C, Marano M, Pirozzi N. Monitoring of intrathoracic volemia and cardiac output in critically ill children. Minerva Anestesiol. 2003 Dec;69(12):907-18. English, Italian. PMID 14743122
- [Background] Cecchetti C, Lubrano R, Cristaldi S, Stoppa F, Barbieri MA, Elli M, Masciangelo R, Perrotta D, Travasso E, Raggi C, Marano M, Pirozzi N. Relationship between global end-diastolic volume and cardiac output in critically ill infants and children. Crit Care Med. 2008 Mar;36(3):928-32. doi: 10.1097/CCM.0B013E31816536F7. PMID 18431282
- [Background] Durand P, Chevret L, Essouri S, Haas V, Devictor D. Respiratory variations in aortic blood flow predict fluid responsiveness in ventilated children. Intensive Care Med. 2008 May;34(5):888-94. doi: 10.1007/s00134-008-1021-z. Epub 2008 Feb 8. PMID 18259726
- [Background] Haque IU, Zaritsky AL. Analysis of the evidence for the lower limit of systolic and mean arterial pressure in children. Pediatr Crit Care Med. 2007 Mar;8(2):138-44. doi: 10.1097/01.PCC.0000257039.32593.DC. PMID 17273118
- [Background] Brierley J, Peters MJ. Distinct hemodynamic patterns of septic shock at presentation to pediatric intensive care. Pediatrics. 2008 Oct;122(4):752-9. doi: 10.1542/peds.2007-1979. PMID 18829798
- [Background] Slater A, Shann F, Pearson G; Paediatric Index of Mortality (PIM) Study Group. PIM2: a revised version of the Paediatric Index of Mortality. Intensive Care Med. 2003 Feb;29(2):278-85. doi: 10.1007/s00134-002-1601-2. Epub 2003 Jan 23. PMID 12541154